CLINICAL TRIAL: NCT03063294
Title: Improving PACT Coordination Across Settings and Services (QUE 15-276)
Brief Title: Coordination Toolkit and Coaching Project
Acronym: CTAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-014
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Results first posted 2020-12-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Coordination, Administrative
Keywords: Coordination, Administrative; Coaching; Primary Care; Quality Improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toolkit only (Active Comparator): Clinics in this arm are given access to an online care coordination toolkit.
  Interventions: Other: Online Toolkit
- Toolkit plus coaching (Experimental): Clinics in this arm are given access to an online care coordination toolkit plus quality improvement support from a distance-based coach.
  Interventions: Other: Online Toolkit; Other: Distance-based coaching

INTERVENTIONS:
Other: Online Toolkit — The online toolkit provides a set of tools that clinics can use to improve their care coordination processes.
Other: Distance-based coaching — The distance-based coach supports included clinics in carrying out a quality improvement project focused on care coordination, either using the online toolkit or other resources determined by the clinic.
  Arms: Toolkit plus coaching

SUMMARY:
The Coordination Toolkit and Coaching (CTAC) project aims to disseminate strategies for coordination of care for high-risk Veterans via an online toolkit, while evaluating the benefits of adding a distance-coaching strategy to assist sites with deploying the toolkit's tools. The project's focus is on care coordination across outpatient settings.

This multi-site project provides: 1) An online toolkit to support better care coordination for vulnerable patients visiting primary care, 2) Random assignment of participating clinics to either a toolkit or a combined toolkit/distance coaching strategy, and 3) A quality improvement approach with "plan-do-study-act" cycles of improvement, designed to support clinics in a locally initiated effort.

The project is recruiting clinics with the goal of improving Veteran experience of care (as measured by a survey called the Hassles Scale).

DETAILED DESCRIPTION:
Background: High-risk Veterans are defined as individuals who are at increased risk for poor clinical outcomes and higher use of unplanned health services relative to their non-high-risk counterparts. These Veterans typically have multiple chronic health problems and are vulnerable to gaps in care due to impaired physical, psychological, and/or social functioning. Despite efforts to integrate care through VA's Patient Aligned Care Teams (PACT) in primary care, deficits in care coordination persist. In VA, most high-risk Veterans are managed in primary care rather than a specialty service. PACT was expected to improve care coordination by creating the care manager role for the PACT teamlet nurse. However, there have been significant challenges in implementing the care manager role as intended. Many of the care coordination challenges involve the "medical neighborhood" outside of PACT.

To improve the quality of care coordination in outpatient care and also develop better methods for spreading innovations, the Coordination Toolkit and Coaching project was funded by VA's Quality Enhancement Research Initiative (QUERI). This project develops and pilots an online toolkit and distance-based coaching process, and then compares the effectiveness of the toolkit alone to the combination of the toolkit plus distance coaching for improving VA patients' experience of care. Both toolkit and combined toolkit/coaching strategies have been used individually in VA quality improvement initiatives, and each strategy has been compared individually to other alternatives. However, to the investigators' knowledge, these strategies have not formally been compared head-to-head.

Additional Outcome Information: The project's primary outcome is a measure of patient experience, the Health System Hassles Scale. This 16-item scale asks patients questions such as whether their medications are being refilled on time, whether they were given information about why they were referred to a specialist, whether there has been poor communication between different doctors or clinics, or whether there have been disagreements between doctors about the patient's diagnosis or the best treatment for the patient.

Sample Size Calculations: The sample size calculation for this study is based on a simple presumption of a difference-in-differences analysis (across the two time points) for the comparison of the two implementation strategies. The primary outcome is the Health System Hassles Scale. The investigators assume 12 clinics in the study (6 per study group), which will be viewed as clusters in order to evaluate the sample size. Since the number of patients per cluster may vary, the investigators assume a coefficient of variation of cluster sizes of about 0.9. With an effect size of 0.3 standard deviations (which is considered to be a small to medium effect size in Cohen's terminology) for the difference-in-difference analysis and an intra-cluster correlation of 0.023 (based on preliminary evaluation of prior data), then with 80% power and two-sided 5% significance level, 149 patients per clinic are needed for a total of 1788 patients (evenly divided between the two groups).

Statistical Analysis Plan: The primary endpoint of the Health System Hassles Scale will be compared between the two implementation groups (toolkit and combined toolkit/coaching) using a difference-in-differences (between the two time points: baseline and 12 months) analysis adjusted for the clustering by clinic. This analysis will be performed initially with a general linear model using the between time point difference as the dependent variable and study group as the independent variable, with clinic as the clustering variable (and, thus, using an appropriately chosen variance-covariance matrix). A further adjustment model may incorporate appropriate covariates including patient-level factors, such as gender, age, and use of non-VA care.

ELIGIBILITY:
Inclusion Criteria:

* VA primary care clinic
* Clinic's facility director must sign a letter of endorsement in support of patients being surveyed about their experience of care
* Identify a clinic champion to serve as point of contact
* Clinic champion has adequate release time to take on a new quality improvement project

Exclusion Criteria:

* Insufficient number of patients to obtain adequate sample size for primary outcome measure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Avram Ganz, MD PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olmos-Ochoa TT, Fenwick KM, Ganz DA, Chawla N, Penney LS, Barnard JM, Miake-Lye IM, Hamilton AB, Finley EP. Reflective writing: a tool to support continuous learning and improved effectiveness in implementation facilitators. Implement Sci Commun. 2021 Sep 3;2(1):98. doi: 10.1186/s43058-021-00203-z. PMID 34479654
- [Derived] Penney LS, Bharath PS, Miake-Lye I, Leng M, Olmos-Ochoa TT, Finley EP, Chawla N, Barnard JM, Ganz DA. Toolkit and distance coaching strategies: a mixed methods evaluation of a trial to implement care coordination quality improvement projects in primary care. BMC Health Serv Res. 2021 Aug 14;21(1):817. doi: 10.1186/s12913-021-06850-1. PMID 34391443
- [Derived] Olmos-Ochoa TT, Ganz DA, Barnard JM, Penney L, Finley EP, Hamilton AB, Chawla N. Sustaining implementation facilitation: a model for facilitator resilience. Implement Sci Commun. 2021 Jun 21;2(1):65. doi: 10.1186/s43058-021-00171-4. PMID 34154670
- [Derived] Noel PH, Barnard JM, Leng M, Penney LS, Bharath PS, Olmos-Ochoa TT, Chawla N, Rose DE, Stockdale SE, Simon A, Lee ML, Finley EP, Rubenstein LV, Ganz DA. The Coordination Toolkit and Coaching Project: Cluster-Randomized Quality Improvement Initiative to Improve Patient Experience of Care Coordination. J Gen Intern Med. 2022 Jan;37(1):95-103. doi: 10.1007/s11606-021-06926-y. Epub 2021 Jun 9. PMID 34109545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited and enrolled VA primary care clinics from October 2016 to June 2018 using a multi-pronged approach, including teleconference presentations and direct outreach to regional and national leadership. Enrolled clinics participated in a 12-month quality improvement project.
Pre-assignment Details: Patient survey data were collected cross-sectionally at baseline and 12-months' follow-up to measure clinic outcomes. For the primary outcome (Health Care System Hassles Scale), both baseline and follow-up data are presented in the "outcomes" section; the primary measure of effectiveness depends on the change in outcome from baseline to follow-up.
Units Other Than Participants: Primary care clinics
Period: Overall Study
Arm/Group | Toolkit Only | Toolkit Plus Coaching
Started (The terminology of "started" applies only to primary care clinics here (only clinics were followed longitudinally). At each clinic, a cross-sectional survey of participants took place at baseline (N=2484), and then a separate cross-sectional survey with a new sample of participants took place at follow-up (N=2481). Since it is incorrect to use the terminology of "started" with respect to participants, we provide the total (baseline plus follow-up) participant sample size (2484+2481=4965).) | 2463; 6 Primary care clinics (2463 equals the sum of 1241 cross-sectional survey respondents at baseline and 1222 at follow-up.) | 2502; 6 Primary care clinics (2502 equals the sum of 1243 cross-sectional survey respondents at baseline and 1259 at follow-up.)
Completed (The terminology of "completed" applies only to primary care clinics here (only clinics were followed longitudinally). At each clinic, a cross-sectional survey of participants took place at baseline (N=2484), and then a separate cross-sectional survey with a new sample of participants took place at follow-up (N=2481). Since it is incorrect to use the terminology of "completed" with respect to participants, we provide the total (baseline plus follow-up) participant sample size (2484+2481=4965).) | 2463; 6 Primary care clinics (2463 equals the sum of 1241 cross-sectional survey respondents at baseline and 1222 at follow-up.) | 2502; 6 Primary care clinics (2502 equals the sum of 1243 cross-sectional survey respondents at baseline and 1259 at follow-up.)
Not Completed | 0; 0 Primary care clinics | 0; 0 Primary care clinics

BASELINE CHARACTERISTICS:
Population: Baseline participant data attributed to analyzed units (i.e., the 12 primary care clinics) come from 2484 clinic participants who responded to a cross-sectional baseline survey at the 12 clinics. Of these individuals, 40 reported receiving no VA care (the clinics being analyzed are part of the VA) in the past 12 months, so they were excluded from further analysis. Data on the remaining 2444 respondents are presented here.
Units Other Than Participants: Primary care clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Toolkit Only | Toolkit Plus Coaching | Total
Number analyzed (Participants) | 1223 | 1221 | 2444
Number analyzed (Primary care clinics) | 6 | 6 | 12
Age, Customized [Count of Participants; unit: Participants]
  Age: 65 or older | 712 | 751 | 1463
  Age: Less than 65 | 508 | 463 | 971
  Age: Unknown | 3 | 7 | 10
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 1036 | 1030 | 2066
  Gender: Female | 180 | 181 | 361
  Gender: Other | 1 | 2 | 3
  Gender: Unknown | 6 | 8 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Non-Hispanic White | 704 | 684 | 1388
  Race/ethnicity: Black or African-American | 137 | 142 | 279
  Race/ethnicity: Hispanic | 142 | 182 | 324
  Race/ethnicity: Asian or Asian-American | 74 | 43 | 117
  Race/ethnicity: Other minority | 27 | 13 | 40
  Race/ethnicity: Multi-race/ethnicity | 66 | 74 | 140
  Race/ethnicity: Unknown race/ethnicity | 73 | 83 | 156

OUTCOME MEASURES:

1. Primary Outcome: Health Care System Hassles Scale
Description: The primary outcome was the 16-item Health Care System Hassles Scale. Recognized as a measure of care coordination, the Hassles questionnaire lists problems that patients may encounter with their general healthcare, as opposed to their care experience with one specific visit or provider. The questionnaire prompts patients to indicate how much situations such as "lack of information about why you've been referred to a specialist" have been a problem, using a 5-point scale ranging from 0 -4. Ratings were dichotomized (0 = "Not a problem at all" vs. 1 = any level of problem indicated) and summed to yield a hassles count ranging from 0 to 16, with higher scores indicating more hassles.
Time Frame: Baseline and 12 months' follow-up
Population: These data derive from two cross-sectional participant surveys at separate (i.e., baseline and follow-up) timepoints. The numbers of participants shown here exceed the numbers presented in the Baseline module because respondents from the surveys are two separate (i.e., independent) samples of participants. Sample sizes for each arm are smaller than reported in the participant flow module because not all survey responses received had valid primary outcome data for analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Units Other Than Participants: Primary care clinics
Arm/Group | Toolkit Only | Toolkit Plus Coaching
Number analyzed (Participants) | 2337 | 2359
Number analyzed (Primary care clinics) | 6 | 6
units on a scale
  Baseline: number analyzed (Participants) | 1179 | 1174
  Baseline | 5.20 [4.95 to 5.46] | 4.71 [4.47 to 4.96]
  12-month Follow-up: number analyzed (Participants) | 1158 | 1185
  12-month Follow-up | 4.78 [4.53 to 5.04] | 4.30 [4.04 to 4.56]
Statistical Analysis 1: Comparison: Toolkit Only; Zero-inflated negative binomial regression was used to obtain predicted mean Hassles scale scores for the "toolkit only" clinics and "toolkit plus coaching" clinics at baseline and follow-up, adjusting for study design and characteristics of survey respondents. The difference-in-difference was then computed as described below, under "method of estimation." Bootstrap resampling was used to calculate the 95% confidence intervals around the predicted means and the difference-in-difference; Test type: Superiority; Difference in Difference = 0.02, 95% CI 2-sided [-0.47 to 0.50] — The difference in difference equals the "follow-up minus baseline" change in Hassles scale results for the "toolkit plus coaching" clinics, minus the "follow-up minus baseline" change in the Hassles scale results for the "toolkit only" clinics

ADVERSE EVENTS:
Time Frame: Not applicable (no adverse event data were collected because the unit of randomization and analysis was the primary care clinic).
Description: Although data were collected for this project from patients served by the clinics using a serial cross-sectional design (in order to determine outcomes for each of the clinics at baseline and follow-up), the patients from whom survey data were collected were not human subjects (this project was determined to be non-research by the VA Greater Los Angeles Healthcare System's Institutional Review Board). Thus, patients were not followed longitudinally and no adverse event data were collected.
Arm/Group | Toolkit Only | Toolkit Plus Coaching
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT03063294/Prot_SAP_000.pdf